CLINICAL TRIAL: NCT00215189
Title: Evaluation of a Health Promotion Intervention for Persons With Mental Illness
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Endowment for Health (Unknown); Robert Wood Johnson Foundation (Other)
Responsible Party: Stephen J. Bartels, MD MS, Dartmouth Medical School
Other Study IDs: IS200406
Record Dates: First submitted 2005-09-15; First posted 2005-09-22 (Estimated); Last update posted 2009-09-23 (Estimated); Status verified 2009-09

CONDITIONS: Mental Illness
Keywords: health; mental illness; fitness
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: In SHAPE (Pilot Health Promotion Intervention)

SUMMARY:
This pilot study evaluates an individualized health promotion program for people with mental illness receiving services at a mental health center in Keene, NH. The study will test the following hypotheses:

Hypothesis 1: Compared to baseline (pre-study) levels, participants in the In SHAPE program will demonstrate increased physical activity as indicated by self-report and observed measures.

Hypothesis 2: Compared to baseline (pre-study) levels, participants in the In SHAPE program will demonstrate improved fitness and health status as indicated by greater capacity on the 6-minute walk test, one mile walk test, weight and body composition, and flexibility indexes.

The following secondary (exploratory) hypotheses will be considered:

Compared to baseline (pre-study) levels, participants in the In SHAPE program will demonstrate improved subjective health status, quality of life, mood, and self-efficacy. In addition, participants will demonstrate improved cardiovascular fitness as indicated by lower pulse rate and blood pressure.

DETAILED DESCRIPTION:
The In SHAPE program aims to improve the physical fitness and health of persons with mental illness. Participants in the program are assigned a health mentor who assesses individual lifestyle habits and health status, identifies goals for lifestyle change, and serves as a motivator and physical trainer. The individualized components of the In SHAPE program are supplemented with group-level positive reinforcement and motivational incentives. This evaluation project systematically evaluates the In SHAPE health promotion intervention.

ELIGIBILITY:
Inclusion Criteria:

Age 18 or older, and enrolled in the In SHAPE program. Mental illness Receiving mental health services for 3 months or longer Voluntary informed consent or guardian consent Signed letter of permission to participate by a physician for individuals with a history of a medical illness or indications of health problems during the evaluation -

Exclusion Criteria:

Inability to give informed, voluntary consent. Primary diagnosis of dementia or a diagnosis of a psychiatric disorder secondary to a medical condition.

Co-morbid dementia as indicated by an MMSE score <20. Exclusion for eligibility as determined by the participant's physician due to medical contraindications (e.g., recent myocardial infarction, stroke (thrombotic or embolic), uncontrolled insulin-dependent diabetes).

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community Mental Health Center
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2004-08; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Bartels, MD, Principal Investigator — Professor in Psychiatry, Dartmouth Medical School
Locations (1):
- Monadnock Family Services, Keene, New Hampshire, United States